CLINICAL TRIAL: NCT02883218
Title: Dynamic Alterations of Th2/Th1 With New Onset of Community-acquired Severe Sepsis
Brief Title: Dynamic Alterations of Th2/Th1 With New Onset of Community-acquired Severe Sepsis Patients
Status: Completed | Type: Observational
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Doctor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: 2014ZDSYLL087.0
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Sepsis
Keywords: immunosuppression; community-acquired sepsis; mortality
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Comunity-acquired severe sepsis patients: Patients with new-onset community-acquired severe sepsis within 24h without confounding factors in immune status
- Non-severe sepsis patients: Patients between 18 and 90 years of age and be admitted to the ICU without a diagnosis of severe sepsis.
- Healthy controls: Heathy vonlunteers between 18 and 90 years of age.

SUMMARY:
To evaluate the dynamic alterations of Th2/Th1 for the prediction of clinical immunity and how it was related to 28 day-prognosis and ICU-acquired infections among critically ill patients of community-acquired severe sepsis with new onset.

ELIGIBILITY:
For community-acquired severe sepsis group:

Inclusion Criteria:

* at least 18 years of age and no more than 90 years of age
* sepsis was defined according to consensus criteria
* diagnosis of sepsis and complicatied with organ dysfunction no longer than 48 h
* provided written informed consent.

Exclusion Criteria:

* diagnosis of hematological,immunological disease or cancer
* treatment with chemotherapy agents or corticosteroids within 6 months prior to or during the hospitalization

For non-severe sepsis ICU control group:

Inclusion Criteria:

* at least 18 years of age and no more than 90 years of age
* without diagnosis of sepsis and admitted to ICU
* provided written informed consent.

Exclusion Criteria:

* diagnosis of hematological,immunological disease or cancer
* treatment with chemotherapy agents or corticosteroids within 6 months prior to or during the hospitalization

For healthy control group:

Inclusion Criteria:

* at least 18 years of age and no more than 90 years of age
* provided written informed consent.

Exclusion Criteria:

* diagnosis of hematological,immunological disease or cancer
* treatment with chemotherapy agents or corticosteroids within 6 months prior to enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enroll patients with community-acquired severe sepsis and then the patients admitted to ICU without the diagnosis of severe sepsis as ICU control group, and the heathy volunteers as healthy control group.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Th2/Th1 upon enrollment | Day 0 after enrollment for community-acquired severe sepsis group and Day 0 after enrollment for the non-severe sepsis patients and heathy control group
  The blood samples were collected for T helper 1 cells and T helper 2 cells populations measured by flow cytometry. All groups are needed.
Th2/Th1 on Day 3 | Day 3 after enrollment for community-acquired severe sepsis group
  populations measured by flow cytometry. Only community-acquired severe sepsis group is needed.
Th2/Th1 on Day 7 | Day 7 after enrollment for community-acquired severe sepsis group
  populations measured by flow cytometry. Only community-acquired severe sepsis group is needed.

SECONDARY OUTCOMES:
28-day mortality for community-acquired severe sepsis group | 28-day
ICU-acquired infection for community-acquired severe sepsis group | 28-day

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xue M, Xie J, Liu L, Huang Y, Guo F, Xu J, Yang Y, Qiu H. Early and dynamic alterations of Th2/Th1 in previously immunocompetent patients with community-acquired severe sepsis: a prospective observational study. J Transl Med. 2019 Feb 27;17(1):57. doi: 10.1186/s12967-019-1811-9. PMID 30813927